CLINICAL TRIAL: NCT06742268
Title: A Multi-center, Open-label, Controlled Extension Study to Evaluate the Rebound Effect and Long-term Safety of Software SAT-001 for the Inhibition of Myopia Progression and Treatment in Pediatric Patients With Myopia
Brief Title: Extension Study on Safety and Rebound Effect of SAT-001 for Myopia in Children
Status: Recruiting | Type: Observational
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAT001-KP-003
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Myopia
Keywords: Myopia; Rebound effect; SaMD
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Spectacles with Cessation of SAT-001 Use: This group consists of pediatric participants who were previously assigned to receive SAT-001 along with single vision spectacles as part of the SAT-001 confirmatory trial (SAT-001-KP-002). In the extension phase, these participants will continue wearing single vision spectacles, but will no longer receive SAT-001 treatment. The aim is to monitor rebound myopia and long-term safety after the completion of the initial trial, focusing on any changes in refractive error and axial length, as well as any adverse effects associated with the cessation of SAT-001 use.
  Interventions: Other: Single vision spectacles
- Arm 2: Continued Spectacles Only: This group consists of pediatric participants who were assigned to the control group during the SAT-001 confirmatory trial and received only single vision spectacles. In the extension phase, they will continue wearing spectacles to assess rebound myopia and long-term safety, without the addition of SAT-001 treatment.
  Interventions: Other: Single vision spectacles

INTERVENTIONS:
Other: Single vision spectacles — Other interventions for myopia treatment, except for glasses, will not be provided.

SUMMARY:
The objective of this clinical trial is to collect data on the rebound effect and long-term safety of SAT-001, a Software as a Medical Device (SaMD) under development for the inhibition and treatment of myopia progression in pediatric patients.

DETAILED DESCRIPTION:
Myopia treatments to date have included both pharmacological and non-pharmacological approaches, with some studies showing effects in reducing myopia progression. However, previous research has also identified a rebound effect, where myopia progresses rapidly after treatment cessation during follow-up. Since myopia progression in children often continues for more than two years, this rebound effect could be a critical factor in determining treatment strategies for pediatric myopia.

This multi-center, open-label, controlled observational study is an extension of a previous confirmatory trial (SAT-001-KP-002) that evaluated SAT-001, a Software as a Medical Device (SaMD) designed to slow myopia progression in pediatric patients. The current study aims to assess the rebound effect and long-term safety of SAT-001 in participants who completed the previous trial, and to collect additional data on rebound myopia and long-term safety outcomes following the completion of the initial trial. A total of 40 participants, aged 5 to less than 9 years, from both the treatment and control groups of the prior study will be followed for 6 months after completing the original trial. Participants from the previous trial who had less than 70% compliance will be excluded from this study. Both groups will continue wearing spectacles, the conventional treatment for myopia, during the extension phase. The primary endpoint is the change in cycloplegic spherical equivalent refractive error (SER) from baseline to 24 weeks, while secondary endpoints include changes in SER at 12 weeks and changes in axial length at 12 and 24 weeks compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the previous clinical trial (SAT001-KP-002), and their legal guardians who agree to participate in this extension study and are willing to provide the signed informed consent after receiving and comprehending the explanation of the description of this clinical trial (subject under 6 can make a mark for agreement after full information and understanding)

Exclusion Criteria:

* Participants in the study group of the previous clinical trial (SAT001-KP-002) with a compliance rate of less than 70% (overall compliance throughout the study period).
* Other reasons for participation in the trial at the discretion of the investigator

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children aged 5 to 8 years at the time of their participation in the previous confirmatory trial (SAT-001-KP-002), who are continuing in the extension study. Participants will remain in their original groups (study or control group) with no new randomization.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
change in spherical equivalent refractive error | baseline, 24 weeks
  change in spherical equivalent refractive error at 24 weeks from baseline

SECONDARY OUTCOMES:
change in spherical equivalent refractive error | Baseline, 12 weeks, 24 weeks
  change in spherical equivalent refractive error at 12- and 24-week from baseline
change in axial length | Baseline, 12 weeks, 24 weeks
  change in axial length at 12-week and 24-week from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paik, MD, Principal Investigator — Gachon University Gil Medical Center; Lee, MD, Principal Investigator — Seoul Asan Medical Center; Han, MD, Principal Investigator — Kangbuk Samsung Hospital; Kim, MD, Principal Investigator — HanGil Eye Hospital; Kim, MD, Principal Investigator — Chung-Ang University Gwang Myeong Hospital; Park, MD, Principal Investigator — Daegu Fatima Hospital; Rhiu, MD, Principal Investigator — Hallym University Dongtan Sacred Heart Hospital
Locations (5):
- South Korea (5):
  - Kangbuk Samsung Hospital, Seoul, Choose One...
  - Seoul Asan Medical Center, Seoul, Choose One...
  - Hallym University Dongtan Sacred heart Hospital, Hwaseong-si, Gyeonggi-do
  - Chung-Ang University Gwang Myeong Hospital, Gwangmyeong
  - Gachon University Gil Medical Center, Incheon

IPD SHARING:
Plan to Share IPD: No